CLINICAL TRIAL: NCT06900764
Title: A Study to Evaluate the Safety and Efficacy of CAR-T Cells in Subjects With Systemic Lupus Erythematosus (SLE)
Brief Title: A Study of CAR-T Cells in Subjects With Systemic Lupus Erythematosus
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Qiubai Li, Director of the Department of Rheumatology and Immunology, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AID04-01
Record Dates: First submitted 2025-03-23; First posted 2025-03-28 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Systemic Lupus Erythematosus (SLE)
Keywords: SLE; Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Immunotherapy, Adoptive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CAR-T treatment (Experimental)
  Interventions: Drug: CAR-T cell

INTERVENTIONS:
Drug: CAR-T cell — CAR-T cell

SUMMARY:
The purpose of this study is to assess the safety and efficacy of CAR-T cell therapy in Subjects with SLE.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, between 18 and 65 years old;
* Diagnosed with SLE according to 2019 EULAR/ACR SLE classifications;
* Positivity for ANA (titer≥1:80), and/or anti-dsDNA, and/or anti-Smith antibody at screening;
* SLEDAI-2K≥8 points (with a clinical SLEDAI-2K≥6 points) ;
* Patients who have used stable standard treatment regimen for at least 6 months in their medical history before screening, and their condition is still active for at least 2 months before screening.
* Good organ functions;
* Voluntary participates this trial and can comprehend and sign ICF.

Exclusion Criteria:

* Had or has active malignancy;
* Had been subjected to treatment by CD19 targeted therapy or CAR-T therapy or any gene therapy;
* Combined with other autoimmune disease that needs treatment;
* Pregnant or lactating women;
* Has other factors that deemed not suitable by investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-10-10 (Estimated); Primary Completion 2027-11-15 (Estimated); Study Completion 2027-12-20 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity | 0~28 day after treatment
Frequency of AEs, SAEs | 0 day to 24 months after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Wuhan Union Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No